CLINICAL TRIAL: NCT06810999
Title: From Fear to Purpose ACT Protocol: Testing Indirect, Transdiagnostic Implications of Death Anxiety Over Depression and Anxiety. A Randomized Placebo Controlled Trial.
Brief Title: From Fear to Purpose ACT Protocol. Implications of Death Anxiety in Depression and Anxiety Symptoms.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Roxana Cardos, PhD, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 816/22.01.2025
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Death Anxiety; Depression; Anxiety
Keywords: death anxiety; depression; anxiety; transdiagnostic; indirect intervention; rct
MeSH Terms: conditions — Necrophobia; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): This arm is the experimental group which will receive the intervention. The intervention is a one session From Fear to Purpose ACT Protocol, which is built on Acceptance and Commitment Therapy (ACT) strategies, focused on identifying and committing to personal values.
  Interventions: Other: From Fear to Purpose (Acceptance and Commitment Therapy)
- Placebo Group (Placebo Comparator): This arm is the placebo group, which will be undergoing a group-based attentional control intervention.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: From Fear to Purpose (Acceptance and Commitment Therapy) — The From Fear to Purpose ACT Protocol is based on Acceptance and Commitment Therapy (ACT) strategies, build around identifying and committing to personal values. The intervention will be group-based (90 minutes session).
  Arms: Experimental Group
Other: Placebo — The placebo condition consists of a group-based attentional control intervention.
  Arms: Placebo Group

SUMMARY:
The main purpose of this placebo controlled trial is to test the efficacy of a one-session From Fear to Purpose ACT intervention in reducing self-reported death anxiety levels. Another objective of this study is to investigate whether reductions in death anxiety levels are associated with reductions in depression and anxiety levels, thus testing if death anxiety is a transdiagnostic factor involved in psychopathology.

DETAILED DESCRIPTION:
This is a placebo controlled trial where the main objective is to test if the one-session From Fear to Purpose ACT intervention is effective in reducing self-reported death anxiety levels. A secondary objective is to investigate whether reductions in death anxiety levels are associated with reductions in depression and anxiety levels, thus testing if death anxiety is a transdiagnostic factor involved in psychopathology.

Participants will be selected based on death anxiety levels (moderate-high scores) and depression and anxiety symptoms (subclinical levels). Minors, people with suicidal ideation, people with current psychological/psychiatric diagnosis (excepting depression or anxiety diagnosis), people in active psychological/psychiatric treatment will be excluded. Recruited participants will be randomized into two groups: the experimental group (will receive the From Fear to Purpose ACT intervention) and the placebo group. The placebo condition will be undergoing a group-based attentional control activity. Participants will be blinded to the study condition.

The From Fear to Purpose intervention protocol is based on Acceptance and Commitment Therapy (ACT) strategies, build around identifying and committing to personal values. The intervention will be group-based (90 minutes session). The intervention will be administered by experienced psychotherapists.

The primary outcome is death anxiety, while secondary outcomes are depression and anxiety symptoms, well-being, psychological flexibility, experiential avoidance and valued living.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-high levels of death anxiety (score > or = 55) AND
* Subclinical levels of depression (score > or = 9) AND/OR
* Subclinical levels of anxiety (score > or = 9)

Exclusion Criteria:

* Minors
* Suicidal ideation
* Current psychological/psychiatric diagnosis (except depression or anxiety diagnosis)
* Active psychological/psychiatric treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Death Anxiety score to the follow-up moment (6 weeks duration) | From enrolment to follow-up (6 weeks time frame)
  Death anxiety measured with Death Anxiety Beliefs and Behaviours Scale (Menzies, Sharpe, Dar-Nimrod, 2022).
  Scores range from 18 to 90, with higher scores indicating higher death anxiety levels.

SECONDARY OUTCOMES:
Change from baseline Depression score to the follow-up moment (6 weeks duration) | From enrolment to follow-up (6 weeks time frame)
  Depression measured with Patient Health Questionnaire - 9 (Kroenke, 1999). Scores range from 0 to 27 with higher scores indicating more severe depression symptoms.
Change from baseline Anxiety score to the follow-up moment (6 weeks duration | From enrolment to follow-up (6 weeks time frame)
  Anxiety measured with Generalized Anxiety Disorder - 7 (Spitzer, 2006). Scores range from 0 to 27, with higher scores indicating more severe anxiety symptoms.
Change from baseline Well-being score to the follow-up moment (6 weeks duration) | From enrolment to follow-up (6 weeks time frame)
  Distress measured with The World Health Organization-Five Well-Being Index (WHO-5; WHO, 2024). Scores range from 0 to 25 with higher scores indicating better well-being.
Change from baseline Psychological Flexibility to the follow-up moment (6 weeks duration) | From enrolment to follow-up (6 weeks time frame)
  Psychological Flexibility measured with Comprehensive assessment of Acceptance and Commitment Therapy processes (CompACT) (Francis, 2016). Scores range from 0 to 138 with higher scores indicating better psychological flexibility.
Change from baseline Experiential Avoidance score to the follow-up moment (6 weeks duration | From enrolment to follow-up (6 weeks time frame)
  Experiential Avoidance measured with Brief Experiential Avoidance Questionnare (Gamez, 2011). Scores range from 15 to 90 with higher scores indicating higher experiential avoidance.
Change from baseline Valued Living score to the follow-up moment (6 weeks duration | From enrolment to follow-up (6 weeks time frame)
  Valued Living measured with Valuing Questionnare (Smout, 2014).
  The measure has two subscales:
  1. Progress, where scores range from 0 to 30, higher scores indicating a closer alignment between one's internal values and one's actions.
  2. Obstruction, where scores range from 0 to 30, higher scores indicating more interference with living consistently with one's values.

OTHER OUTCOMES:
Satisfaction with the intervention protocol | One month
  Satisfaction with the intervention protocol measured with Client Satisfaction Questionnaire - 8 (Attkisson, 1982). Measured post intervention and at follow-up for the experimental group.
  Scores range from 8 to 32, higher scores indicating greater satisfaction with the intervention.

IPD SHARING:
Plan to Share IPD: Yes
Will share IPD used in the results of the publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD will be shared after publication with no end date. The Study Protocol will be shared in March 2025 with no end date. The Statistical Analysis Plan will be shared in March 2025 with no end date. The Informed Consent Form will be shared in March 2025 with no end date.